CLINICAL TRIAL: NCT04739254
Title: Magnetocardiography Endocrine Registry
Acronym: MACENDOR
Status: Suspended | Type: Observational
Why Stopped: Resourcing
Sponsor: Genetesis Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1000-4
Record Dates: First submitted 2021-01-27; First posted 2021-02-04 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Endocrine Disorder
Keywords: endocrine disorders; MCG; Cardiovascular disease; ischemia; CardioFlux
MeSH Terms: conditions — Endocrine System Diseases; Cardiovascular Diseases; Ischemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: CardioFlux — Magnetocardiography

SUMMARY:
Endocrine disorders like Type 2 diabetes mellitus (T2DM) represent complex cardiometabolic disease processes affecting approximately 462 million individuals worldwide and is associated with a two- to three-fold increase in cardiovascular mortality. Individuals with T2DM are at an increased risk of developing cardiovascular disease. Research has shown individuals with T2DM and no previous history of coronary artery disease are still at similar risk rates for cardiovascular events as patients with a prior myocardial infarction. The MAgenetoCardiography ENDOcrine Registry (MACENDOR) study is designed to collect CardioFlux scans on a select group of volunteers who are high-risk patients with endocrine disorders. CardioFlux is used as a noninvasive magnetocardiography (MCG) tool that analyzes and records the magnetic fields of the heart to screen volunteers for heart disease. There will be a 12-month duration of the study where we propose to collect screening data from approximately 250 volunteers who present to the Genetesis facility for a 5-minute CardioFlux scan. The volunteers will be contacted at intervals over a 1-year period for follow-up data and may choose whether or not they would like to provide follow-up data or participate in another scan.

ELIGIBILITY:
Inclusion Criteria:

1. ≥ 18 years of age at the time of enrollment
2. Patients deemed at risk for cardiovascular disease from endocrine disorders

Exclusion Criteria:

1. < 18 years of age
2. Patients unable to fit into device
3. Non-ambulatory patients
4. Positive response(s) on CardioFlux Pre-Screening Form
5. Patients with claustrophobia or unable to lie supine for five minutes
6. Pregnant women
7. Poor candidates for follow-up (e.g., no access to phone)
8. Prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are at risk for cardiovascular disease due to endocrine disorders.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2020-12-14 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2030-05-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy statistics | 12 months
  analyzing the accuracy of CardioFlux
Specificity statistics | 12 months
  analyzing the specificity of CardiFlux

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Senagore, M.D., Principal Investigator — Genetesis Inc.
Locations (1):
- Genetesis Facility, Mason, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ogurtsova K, da Rocha Fernandes JD, Huang Y, Linnenkamp U, Guariguata L, Cho NH, Cavan D, Shaw JE, Makaroff LE. IDF Diabetes Atlas: Global estimates for the prevalence of diabetes for 2015 and 2040. Diabetes Res Clin Pract. 2017 Jun;128:40-50. doi: 10.1016/j.diabres.2017.03.024. Epub 2017 Mar 31. PMID 28437734
- [Background] Rao Kondapally Seshasai S, Kaptoge S, Thompson A, Di Angelantonio E, Gao P, Sarwar N, Whincup PH, Mukamal KJ, Gillum RF, Holme I, Njolstad I, Fletcher A, Nilsson P, Lewington S, Collins R, Gudnason V, Thompson SG, Sattar N, Selvin E, Hu FB, Danesh J; Emerging Risk Factors Collaboration. Diabetes mellitus, fasting glucose, and risk of cause-specific death. N Engl J Med. 2011 Mar 3;364(9):829-841. doi: 10.1056/NEJMoa1008862. PMID 21366474
- [Background] Emerging Risk Factors Collaboration; Di Angelantonio E, Kaptoge S, Wormser D, Willeit P, Butterworth AS, Bansal N, O'Keeffe LM, Gao P, Wood AM, Burgess S, Freitag DF, Pennells L, Peters SA, Hart CL, Haheim LL, Gillum RF, Nordestgaard BG, Psaty BM, Yeap BB, Knuiman MW, Nietert PJ, Kauhanen J, Salonen JT, Kuller LH, Simons LA, van der Schouw YT, Barrett-Connor E, Selmer R, Crespo CJ, Rodriguez B, Verschuren WM, Salomaa V, Svardsudd K, van der Harst P, Bjorkelund C, Wilhelmsen L, Wallace RB, Brenner H, Amouyel P, Barr EL, Iso H, Onat A, Trevisan M, D'Agostino RB Sr, Cooper C, Kavousi M, Welin L, Roussel R, Hu FB, Sato S, Davidson KW, Howard BV, Leening MJ, Leening M, Rosengren A, Dorr M, Deeg DJ, Kiechl S, Stehouwer CD, Nissinen A, Giampaoli S, Donfrancesco C, Kromhout D, Price JF, Peters A, Meade TW, Casiglia E, Lawlor DA, Gallacher J, Nagel D, Franco OH, Assmann G, Dagenais GR, Jukema JW, Sundstrom J, Woodward M, Brunner EJ, Khaw KT, Wareham NJ, Whitsel EA, Njolstad I, Hedblad B, Wassertheil-Smoller S, Engstrom G, Rosamond WD, Selvin E, Sattar N, Thompson SG, Danesh J. Association of Cardiometabolic Multimorbidity With Mortality. JAMA. 2015 Jul 7;314(1):52-60. doi: 10.1001/jama.2015.7008. PMID 26151266
- [Background] Tancredi M, Rosengren A, Svensson AM, Kosiborod M, Pivodic A, Gudbjornsdottir S, Wedel H, Clements M, Dahlqvist S, Lind M. Excess Mortality among Persons with Type 2 Diabetes. N Engl J Med. 2015 Oct 29;373(18):1720-32. doi: 10.1056/NEJMoa1504347. PMID 26510021
- [Background] Simmons RK, Griffin SJ, Lauritzen T, Sandbaek A. Effect of screening for type 2 diabetes on risk of cardiovascular disease and mortality: a controlled trial among 139,075 individuals diagnosed with diabetes in Denmark between 2001 and 2009. Diabetologia. 2017 Nov;60(11):2192-2199. doi: 10.1007/s00125-017-4299-y. Epub 2017 Aug 23. PMID 28831539